CLINICAL TRIAL: NCT01434147
Title: Preoperative Induction Chemotherapy in Combination With Bevacizumab Followed by Combined Chemoradiotherapy in Locally Advanced Rectal Cancer With High Risk of Recurrence- Phase II Pilot Study With Preoperative Administration of Capecitabine (Xeloda), Oxaliplatin and Bevacizumab (Avastin) Followed by Capecitabine (Xeloda) Plus Radiotherapy (RTx)
Brief Title: Preoperative Combined Induction Chemotherapy With Capecitabine, Oxaliplatin, Bevacizumab and Radiotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABCSG R05; 2010-024354-11 (EudraCT Number)
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Rectal Cancer
Keywords: locally advanced rectal cancer; preoperative induction chemotherapy chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Bevacizumab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- induction chemotherapy + radiochemotherapy (Experimental): preoperative induction chemotherapy in combination with bevacizumab followed by combined radiochemotherapy with capecitabine induction chemotherapy: starts within 28 days after bioptical diagnosis. All patients are administered with capecitabine (Xeloda®) 1000 mg/m2 bid during 14 days (d1-d14), oxaliplatin 130 mg/m2 and bevacizumab (Avastin®) 7.5 mg/kg body weight on day 1; repetition days 22 and 43 (3 cycles) Combined radiochemotherapy: starts at the earliest one week after concluded third cycle of induction chemotherapy. Radiotherapy takes place on 5 x 5 days (dose: 1.8 Gy; cumulative dose: 45 Gy). For chemotherapy patients are administered with capecitabine (Xeloda®) 825mg/m² bid, on each radiation day during the first 4 weeks of radiochemotherapy.
  Interventions: Drug: preoperative induction chemotherapy in combination with bevacizumab followed by combined radiochemotherapy with capecitabine

INTERVENTIONS:
Drug: preoperative induction chemotherapy in combination with bevacizumab followed by combined radiochemotherapy with capecitabine — Therapy start: Capecitabine 1000mg/ m² bid during 14 days(d1-14), oxaliplatin 130mg/m² and Bevacizumab 7.5mg/kg body weight d1, repetition day 22 and 43 (3 cycles) Radiotherapy: Followed by 5 x 5 days 1.8 Gy after 1 week of concluded 3rd cycle of induction chemotherapy Chemotherapy: Capecitabine 825 mg/m2 bid (on each therapy day of first 4 therapy weeks)
  Other Names: Xeloda (capecitabine); Avastin (bevacizumab); Oxaliplatin

SUMMARY:
Phase II pilot study of a preoperative induction chemotherapy in combination with Bevacizumab followed by combined radiochemotherapy for patients with locally advanced rectal carcinoma

DETAILED DESCRIPTION:
Induction chemotherapy combined with Radio chemotherapy:

Therapy start: within 28 days after bioptical diagnosis capecitabine 1000 mg/m2 bid during 14 days (d1-d14) , oxaliplatin 130 mg/m2 and bevacizumab 7.5 mg/kg body weight d1; repetition day 22 and 43 (3 cycles)

Combined Radiochemotherapy after 1 week of concluded 3rd cycle of induction chemotherapy:

Radiotherapy: 5 x 5 days 1.8 Gy; cumulative dose 45 Gy Chemotherapy: capecitabine 825mg/m² bid, on each radiation day during the first 4 weeks of RCTx

Surgery according to TME-criteria (total mesorectal excision) in compliance of an interruption of min. 14 days after RCTx

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Histologic confirmation of rectal adenocarcinoma stage cT3 (≤ 5mm to the mesorectal fascia)/cT4( primary curative intention)NxM0
* No former chemotherapy, no former radiotherapy of the pelvic, no former tumour resection of a rectal carcinoma
* General condition WHO grade 0-2
* Adequate bone marrow reserve ( leucocytes ≥3 000/μl, thrombocytes ≥100 000/μl)
* Adequate renal function (creatinine ≤ 1,5 mg/dl, creatinine clearance > 50ml/min (Cockcroft and Gault formula))
* Adequate liver function (bilirubin ≤1,5x ULN, GOT and GPT ≤3,5xULN)
* Exclusion of pregnancy for women with childbearing potential (negative pregnancy test urine or serum)
* Female patients with childbearing potential and male patients that are not surgically sterile must be practicing a medically acceptable contraceptive regimen while on study treatment until 3 months after the end of the study (e.g. oral contraceptives, condom, intrauterine device)
* Life expectancy of at least 3 months
* INR and aPTT ≤ 1,5 x LLN
* Provision of signed informed consents before registration

Exclusion Criteria:

* Rectal carcinoma stage cT3 (> 5mm from the mesorectal fascia) all stages <cT3, M1
* Other malignant tumours within the last 5 years except cervical carcinoma in situ and basal cell carcinoma of the skin
* General contraindication or known hypersensitivity against Bevacizumab, Capecitabine and Oxaliplatin
* Not malignant diseases for which treatment with radiotherapy, resection of the rectum and treatment with chemotherapy (Bevacizumab, Capecitabine) is contraindicated: uncontrolled hypertension (systolic > 150 mmHG and/or diastolic > 100 mmHG) or clinically significant (e.g. active) cardiovascular diseases: CVA (cardiovascular accident)/ apoplectic insult (≤ 6 months prior to registration), myocardial infarction (≤ 6 months prior to registration), unstable angina pectoris, CHF(congestive heart failure) with NYHA (New York heart Association) Grade II or higher, cardiac arrhythmia requiring therapy, hepatic diseases, significant neurologic or psychiatric disorders
* Florid, serious infection at registration
* Peripheral neuropathy (NCI CTCAE v 4.0 ≥ grade 1)
* Juridically limited contractual capability, indication of neurological or psychiatric disease which constrains upon investigators opinion the patients capability to adhere to the study routines
* Major surgical procedure within 28 days prior start of the study, open wounds
* Significant traumatic injury, bone fracture, unhealed wounds
* Patients with spinal cord compression or metastases in the central nervous system
* Indication of bleeding diathesis or coagulopathy
* Intake of anticoagulant or thrombolytic agents and/or Aspirin > 325 mg/d within 10 days prior to registration
* Current or recent (within 10 days prior to treatment start) therapy with full dosed anticoagulants. Preventive therapy is allowed.
* Previous thromboembolic or haemorrhagic events within 6 months prior to registration
* Previous abdominal fistulas, gastro-intestinal perforation or intrabdominal abscesses within 6 months prior to registration
* Treatment with another investigational drug within 28 days prior to registration
* Patients with malabsorption syndrome or difficulties in swallowing
* Indication of poor compliance of the patient
* Pregnant or breast-feeding women
* Proteinuria: Dipstick <2+. If the Dipstick is ≥2+ protein has to be estimated in the 24 hours urine. The value should not be higher then 1g/24 hours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
termination of therapy | up to 17 weeks
  before surgery (after conclusion of therapy phase)
occurence of toxicity | up to 18-19 weeks
  until timepoint of discharge of patient

SECONDARY OUTCOMES:
collection of response rate | up to week 18
  T- and N-downstaging, pathological complete remission: measurement at the timepoint of surgery
post-surgery morbidity | after 18-19 weeks
  according to Accordion; measurement at the timepoint of discharge of patient

CONTACTS AND LOCATIONS:
Overall Officials: Dietmar Öfner, MD, Head, Study Chair — Austrian Breast & Colorectal Cancer Study Group; Alexander de Vries, MD, Head, Study Chair — Austrian Breast & Colorectal Cancer Study Group; Wolfgang Eisterer, MD, Study Chair — Austrian Breast & Colorectal Cancer Study Group
Locations (7):
- Austria (7):
  - Hospital BHB St. Veit/Glan, Surgery, Saint Veit A. D. Glan, Carinthia
  - Paracelsus Medical University Salzburg - Oncology, Salzburg, Salzburg
  - Medical University Graz, Oncology, Graz, Styria
  - Medical University Innsbruck, Internal Medicine, Innsbruck, Tyrol
  - Klinikum Wels-Grieskirchen, Wels, Upper Austria
  - Medical University of Vienna, General Hospital, Vienna, Vienna
  - State Hospital Feldkirch, Radiotherapy, Feldkirch, Vorarlberg

REFERENCES:
- [Background] NIH consensus conference. Intravenous immunoglobulin. Prevention and treatment of disease. JAMA. 1990 Dec 26;264(24):3189-93. No abstract available. PMID 2255028
- [Background] Goldberg RM, Sargent DJ, Morton RF, Fuchs CS, Ramanathan RK, Williamson SK, Findlay BP, Pitot HC, Alberts SR. A randomized controlled trial of fluorouracil plus leucovorin, irinotecan, and oxaliplatin combinations in patients with previously untreated metastatic colorectal cancer. J Clin Oncol. 2004 Jan 1;22(1):23-30. doi: 10.1200/JCO.2004.09.046. Epub 2003 Dec 9. PMID 14665611
- [Background] MacFarlane JK, Ryall RD, Heald RJ. Mesorectal excision for rectal cancer. Lancet. 1993 Feb 20;341(8843):457-60. doi: 10.1016/0140-6736(93)90207-w. PMID 8094488
- [Background] Budach et al. Stellenwert der Radio- und Radiochemotherapie beim Rektumkarzinom. Onkologe 1998;4:40-48
- [Background] Kockerling F, Reymond MA, Altendorf-Hofmann A, Dworak O, Hohenberger W. Influence of surgery on metachronous distant metastases and survival in rectal cancer. J Clin Oncol. 1998 Jan;16(1):324-9. doi: 10.1200/JCO.1998.16.1.324. PMID 9440760
- [Background] Valentini V, Aristei C, Glimelius B, Minsky BD, Beets-Tan R, Borras JM, Haustermans K, Maingon P, Overgaard J, Pahlman L, Quirke P, Schmoll HJ, Sebag-Montefiore D, Taylor I, Van Cutsem E, Van de Velde C, Cellini N, Latini P; Scientific Committee. Multidisciplinary Rectal Cancer Management: 2nd European Rectal Cancer Consensus Conference (EURECA-CC2). Radiother Oncol. 2009 Aug;92(2):148-63. doi: 10.1016/j.radonc.2009.06.027. PMID 19595467
- [Background] Tournigand C, Andre T, Achille E, Lledo G, Flesh M, Mery-Mignard D, Quinaux E, Couteau C, Buyse M, Ganem G, Landi B, Colin P, Louvet C, de Gramont A. FOLFIRI followed by FOLFOX6 or the reverse sequence in advanced colorectal cancer: a randomized GERCOR study. J Clin Oncol. 2004 Jan 15;22(2):229-37. doi: 10.1200/JCO.2004.05.113. Epub 2003 Dec 2. PMID 14657227
- [Background] Arkenau HT, Arnold D, Cassidy J, Diaz-Rubio E, Douillard JY, Hochster H, Martoni A, Grothey A, Hinke A, Schmiegel W, Schmoll HJ, Porschen R. Efficacy of oxaliplatin plus capecitabine or infusional fluorouracil/leucovorin in patients with metastatic colorectal cancer: a pooled analysis of randomized trials. J Clin Oncol. 2008 Dec 20;26(36):5910-7. doi: 10.1200/JCO.2008.16.7759. Epub 2008 Nov 17. PMID 19018087
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Kabbinavar FF, Hambleton J, Mass RD, Hurwitz HI, Bergsland E, Sarkar S. Combined analysis of efficacy: the addition of bevacizumab to fluorouracil/leucovorin improves survival for patients with metastatic colorectal cancer. J Clin Oncol. 2005 Jun 1;23(16):3706-12. doi: 10.1200/JCO.2005.00.232. Epub 2005 May 2. PMID 15867200
- [Background] Giantonio BJ, Catalano PJ, Meropol NJ, O'Dwyer PJ, Mitchell EP, Alberts SR, Schwartz MA, Benson AB 3rd; Eastern Cooperative Oncology Group Study E3200. Bevacizumab in combination with oxaliplatin, fluorouracil, and leucovorin (FOLFOX4) for previously treated metastatic colorectal cancer: results from the Eastern Cooperative Oncology Group Study E3200. J Clin Oncol. 2007 Apr 20;25(12):1539-44. doi: 10.1200/JCO.2006.09.6305. PMID 17442997
- [Background] Saltz LB, Clarke S, Diaz-Rubio E, Scheithauer W, Figer A, Wong R, Koski S, Lichinitser M, Yang TS, Rivera F, Couture F, Sirzen F, Cassidy J. Bevacizumab in combination with oxaliplatin-based chemotherapy as first-line therapy in metastatic colorectal cancer: a randomized phase III study. J Clin Oncol. 2008 Apr 20;26(12):2013-9. doi: 10.1200/JCO.2007.14.9930. PMID 18421054
- [Background] Tebutt et al. International randomized phase III study of Capecitabine (Cap), bevacizumab (Bev), and mitomycin C (MMC) in first-line metastatic colorectal cancer (mCRC): Final results of the AGITG MAX trial. Proc ASCO 2010, #3538
- [Background] Willett CG, Boucher Y, di Tomaso E, Duda DG, Munn LL, Tong RT, Chung DC, Sahani DV, Kalva SP, Kozin SV, Mino M, Cohen KS, Scadden DT, Hartford AC, Fischman AJ, Clark JW, Ryan DP, Zhu AX, Blaszkowsky LS, Chen HX, Shellito PC, Lauwers GY, Jain RK. Direct evidence that the VEGF-specific antibody bevacizumab has antivascular effects in human rectal cancer. Nat Med. 2004 Feb;10(2):145-7. doi: 10.1038/nm988. Epub 2004 Jan 25. PMID 14745444
- [Background] Willett CG, Boucher Y, Duda DG, di Tomaso E, Munn LL, Tong RT, Kozin SV, Petit L, Jain RK, Chung DC, Sahani DV, Kalva SP, Cohen KS, Scadden DT, Fischman AJ, Clark JW, Ryan DP, Zhu AX, Blaszkowsky LS, Shellito PC, Mino-Kenudson M, Lauwers GY. Surrogate markers for antiangiogenic therapy and dose-limiting toxicities for bevacizumab with radiation and chemotherapy: continued experience of a phase I trial in rectal cancer patients. J Clin Oncol. 2005 Nov 1;23(31):8136-9. doi: 10.1200/JCO.2005.02.5635. No abstract available. PMID 16258121
- [Background] Strasberg SM, Linehan DC, Hawkins WG. The accordion severity grading system of surgical complications. Ann Surg. 2009 Aug;250(2):177-86. doi: 10.1097/SLA.0b013e3181afde41. PMID 19638919
- [Background] ABCSG; ACO/ASSO; OGC; OGHO; OGP; OGRO; ORG. [Recommendations on the diagnosis and multimodal primary therapy of rectal carcinomas 2004]. Wien Klin Wochenschr. 2005 Feb;117(4):154-71. doi: 10.1007/s00508-005-0323-1. No abstract available. German. PMID 15847197
- [Background] de Gramont A, Tournigand C, Andre T, Larsen AK, Louvet C. Adjuvant therapy for stage II and III colorectal cancer. Semin Oncol. 2007 Apr;34(2 Suppl 1):S37-40. doi: 10.1053/j.seminoncol.2007.01.004. PMID 17449351
- [Background] Twelves C, Wong A, Nowacki MP, Abt M, Burris H 3rd, Carrato A, Cassidy J, Cervantes A, Fagerberg J, Georgoulias V, Husseini F, Jodrell D, Koralewski P, Kroning H, Maroun J, Marschner N, McKendrick J, Pawlicki M, Rosso R, Schuller J, Seitz JF, Stabuc B, Tujakowski J, Van Hazel G, Zaluski J, Scheithauer W. Capecitabine as adjuvant treatment for stage III colon cancer. N Engl J Med. 2005 Jun 30;352(26):2696-704. doi: 10.1056/NEJMoa043116. PMID 15987918
- [Background] Andre T, Boni C, Navarro M, Tabernero J, Hickish T, Topham C, Bonetti A, Clingan P, Bridgewater J, Rivera F, de Gramont A. Improved overall survival with oxaliplatin, fluorouracil, and leucovorin as adjuvant treatment in stage II or III colon cancer in the MOSAIC trial. J Clin Oncol. 2009 Jul 1;27(19):3109-16. doi: 10.1200/JCO.2008.20.6771. Epub 2009 May 18. PMID 19451431
- [Background] Kuebler JP, Wieand HS, O'Connell MJ, Smith RE, Colangelo LH, Yothers G, Petrelli NJ, Findlay MP, Seay TE, Atkins JN, Zapas JL, Goodwin JW, Fehrenbacher L, Ramanathan RK, Conley BA, Flynn PJ, Soori G, Colman LK, Levine EA, Lanier KS, Wolmark N. Oxaliplatin combined with weekly bolus fluorouracil and leucovorin as surgical adjuvant chemotherapy for stage II and III colon cancer: results from NSABP C-07. J Clin Oncol. 2007 Jun 1;25(16):2198-204. doi: 10.1200/JCO.2006.08.2974. Epub 2007 Apr 30. PMID 17470851
- [Background] Haller et al. A randomized phase III trial of Capecitabin + oxaliplatin (XELOX) versus bolus 5-FU/LV for stage III colon cancer. ECCO/ESMO 2009, #LBA5.
- [Background] NCCN Clinical Practice guidelines in Oncology (NCCN GuidelinesTM) Rectal cancer version 2.2011. NCCN.org
- [Background] Chau I, Brown G, Cunningham D, Tait D, Wotherspoon A, Norman AR, Tebbutt N, Hill M, Ross PJ, Massey A, Oates J. Neoadjuvant capecitabine and oxaliplatin followed by synchronous chemoradiation and total mesorectal excision in magnetic resonance imaging-defined poor-risk rectal cancer. J Clin Oncol. 2006 Feb 1;24(4):668-74. doi: 10.1200/JCO.2005.04.4875. PMID 16446339
- [Background] Marechal et al. Chemotherapy induction followed by preoperative chemoradiation versus preoperative chemoradiation alone in locally advanced rectal cancer (LARC): A randomized controlled phase II study. Proc ASCO 2010: abstract 3637
- [Background] Fernandez-Martos C, Pericay C, Aparicio J, Salud A, Safont M, Massuti B, Vera R, Escudero P, Maurel J, Marcuello E, Mengual JL, Saigi E, Estevan R, Mira M, Polo S, Hernandez A, Gallen M, Arias F, Serra J, Alonso V. Phase II, randomized study of concomitant chemoradiotherapy followed by surgery and adjuvant capecitabine plus oxaliplatin (CAPOX) compared with induction CAPOX followed by concomitant chemoradiotherapy and surgery in magnetic resonance imaging-defined, locally advanced rectal cancer: Grupo cancer de recto 3 study. J Clin Oncol. 2010 Feb 10;28(5):859-65. doi: 10.1200/JCO.2009.25.8541. Epub 2010 Jan 11. PMID 20065174
- [Background] Dipetrillo T, Pricolo V, Lagares-Garcia J, Vrees M, Klipfel A, Cataldo T, Sikov W, McNulty B, Shipley J, Anderson E, Khurshid H, Oconnor B, Oldenburg NB, Radie-Keane K, Husain S, Safran H. Neoadjuvant bevacizumab, oxaliplatin, 5-fluorouracil, and radiation for rectal cancer. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):124-9. doi: 10.1016/j.ijrobp.2010.08.005. Epub 2010 Oct 13. PMID 20947267
- [Background] Ofner D, Devries AF, Schaberl-Moser R, Greil R, Rabl H, Tschmelitsch J, Zitt M, Kapp KS, Fastner G, Keil F, Eisterer W, Jager R, Offner F, Gnant M, Thaler J; TAKO 05/ABCSG R-02 Trial Investigators. Preoperative oxaliplatin, capecitabine, and external beam radiotherapy in patients with newly diagnosed, primary operable, cT(3)NxM0, low rectal cancer: a phase II study. Strahlenther Onkol. 2011 Feb;187(2):100-7. doi: 10.1007/s00066-010-2182-6. Epub 2011 Jan 21. PMID 21267531
- [Background] Gerard JP, Azria D, Gourgou-Bourgade S, Martel-Laffay I, Hennequin C, Etienne PL, Vendrely V, Francois E, de La Roche G, Bouche O, Mirabel X, Denis B, Mineur L, Berdah JF, Mahe MA, Becouarn Y, Dupuis O, Lledo G, Montoto-Grillot C, Conroy T. Comparison of two neoadjuvant chemoradiotherapy regimens for locally advanced rectal cancer: results of the phase III trial ACCORD 12/0405-Prodige 2. J Clin Oncol. 2010 Apr 1;28(10):1638-44. doi: 10.1200/JCO.2009.25.8376. Epub 2010 Mar 1. PMID 20194850
- [Background] Aschele C, Cionini L, Lonardi S, Pinto C, Cordio S, Rosati G, Artale S, Tagliagambe A, Ambrosini G, Rosetti P, Bonetti A, Negru ME, Tronconi MC, Luppi G, Silvano G, Corsi DC, Bochicchio AM, Chiaulon G, Gallo M, Boni L. Primary tumor response to preoperative chemoradiation with or without oxaliplatin in locally advanced rectal cancer: pathologic results of the STAR-01 randomized phase III trial. J Clin Oncol. 2011 Jul 10;29(20):2773-80. doi: 10.1200/JCO.2010.34.4911. Epub 2011 May 23. PMID 21606427
- [Background] Valentini V, Coco C, Picciocchi A, Morganti AG, Trodella L, Ciabattoni A, Cellini F, Barbaro B, Cogliandolo S, Nuzzo G, Doglietto GB, Ambesi-Impiombato F, Cosimelli M. Does downstaging predict improved outcome after preoperative chemoradiation for extraperitoneal locally advanced rectal cancer? A long-term analysis of 165 patients. Int J Radiat Oncol Biol Phys. 2002 Jul 1;53(3):664-74. doi: 10.1016/s0360-3016(02)02764-5. PMID 12062610
- [Background] Rodel C, Liersch T, Hermann RM, Arnold D, Reese T, Hipp M, Furst A, Schwella N, Bieker M, Hellmich G, Ewald H, Haier J, Lordick F, Flentje M, Sulberg H, Hohenberger W, Sauer R. Multicenter phase II trial of chemoradiation with oxaliplatin for rectal cancer. J Clin Oncol. 2007 Jan 1;25(1):110-7. doi: 10.1200/JCO.2006.08.3675. PMID 17194912
- [Background] Francois Y, Nemoz CJ, Baulieux J, Vignal J, Grandjean JP, Partensky C, Souquet JC, Adeleine P, Gerard JP. Influence of the interval between preoperative radiation therapy and surgery on downstaging and on the rate of sphincter-sparing surgery for rectal cancer: the Lyon R90-01 randomized trial. J Clin Oncol. 1999 Aug;17(8):2396. doi: 10.1200/JCO.1999.17.8.2396. PMID 10561302
- [Background] Lim SB, Choi HS, Jeong SY, Kim DY, Jung KH, Hong YS, Chang HJ, Park JG. Optimal surgery time after preoperative chemoradiotherapy for locally advanced rectal cancers. Ann Surg. 2008 Aug;248(2):243-51. doi: 10.1097/SLA.0b013e31817fc2a0. PMID 18650634
- [Background] S3-Leitlinie "Kolorektales Karzinom, Arbeitsgruppe "Workflow Rektumkarzinom" Zentralbl Chir 2006; 131:285-297
- [Result] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- See also: open studies — http://abcsg.at